CLINICAL TRIAL: NCT01715740
Title: Study of the Effects of Antipruritic Chinese Herbal Medicine on Chronic Urticaria: a Randomized, Double-blind, Placebo-controlled, Phase III Clinical Trial.
Brief Title: Study of the Effects of Chinese Herbal Medicine on Chronic Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, YANG SIEN-HUNG, Director of Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG1B0081
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Urticaria
Keywords: Chinese herbal medicine; Urticaria; Antipruritics; Phase III clinical trial
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — Yi-Gan San

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese herbal medicine (CHM) (Experimental): Subject in CHM group will receive CHM capsules, 8 capsules (4 gm) four times a day, total 16 gm a day, combined with levocetiricine 1PC once a day for 1 month.
  Interventions: Drug: Chinese Herbal Medicine (CHM)
- Control (Placebo Comparator): Subjects in control group will receive the placebo capsules, which has the similar look, smell and taste. The dosage, frequency and duration are the same as CHM group, in which 8 placebo capsule (4gm) 4 times a day, total 16 gm a day, combined with levocetiricine 1PC once a day, for 1 month.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chinese Herbal Medicine (CHM) — Each CHM capsule, weighing 500mg, consists of XFS 250 mg and QSFFT 250 mg.
  Other Names: XFS (Xiao-feng-san):; - Hsiao-feng-san; - yokukansan; - Eliminate Wind Powder; QSFFT (Qin-shang-fang-fen-tang); - Qing-shang-fang-feng-tang
  Arms: Chinese herbal medicine (CHM)
Drug: Placebo — Encapsulated powder with similar taste, color, odor to intervention Chinese herbal medicine
  Arms: Control

SUMMARY:
Urticaria is a common dermatology disease. Urticaria affects nearly 25% of the population at some time in their lives. Recurrent skin itch, insomnia, daily activities limitation greatly affect the quality of life. Some patient with chronic urticaria who had poor response to antihistamine may need second line medication. In United States, up to 54% chronic urticarial patient use oral corticosteroid to control. However, long-term use of oral steroids still needs to consider the impact of its side effects. Therefore, patients may seek for alternative medicine as an adjuvant therapy.

It is still lack large-scale clinical trials in Traditional Chinese Medicine research of chronic urticarial. The aim of this study is to conduct a double-blind, randomized clinical trial to analyze the effectiveness of Chinese medicine in chronic urticaria and its possible mechanisms.

DETAILED DESCRIPTION:
Traditional Chinese medicine has been used widely in Taiwan for several diseases, such as allergic rhinitis, atopic dermatitis. For urticaria,certain antipruritic Chinese herbal medicine, such and Xiao-feng-san (XFS), Qing-shang-fang-fen-tang (QSFFT), have been commonly used in clinical practice, yet no clinical trials have been done to prove the effectiveness.

In this study, a double-blinded, randomized, placebo control trial is designed and total 100 chronic urticaria patients will be enrolled. All subjects will be divided into Chinese herbal medicine (CHM) and placebo control groups, in 1:1 allocation ratio. CHM group will receive capsule of mixture of XFS and QSFFT, 4gm four times a day, total 16 gm in a single day; while control group will receive placebo capsule with similar look, smell, and taste with same scheme. Total 1 month treatment course with 1 month follow-up study course will be done. Changes in symptom severity is the primary outcome, while improvement in sleep disturbance, and serologic marker evolution are the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as idiopathic urticaria at least 6 weeks
* Ages from 18 to 75 years
* Symptom severity must be above 10 points (UAS7 scoring)
* Will to complete questionnaires and take medicine as schedule in this study
* Volunteer for study enrollment and sign inform consent

Exclusion Criteria:

* Other dermatological diseases related to skin pruritus, judged by clinician
* Systemic diseases, such as cancer, renal diseases, liver diseases, autoimmune diseases, and acute infectious diseases. Judged by clinician
* Using oral/injected steroid, leukotriene inhibitors, immuno-suppressant, or other Chinese herbal medicine during one month before enrollment
* Abnormal hemogram, liver or renal function tests in laboratory examination
* Women who are pregnant or are planned to conceive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in symptom severity | Assessment of symptom severity on starting day (day 0), day 7, day 28, day 35 and day 56 for UAS7, and the DLQI on starting day (day 0), day 28 and day 56
  Weekly urticaria activity score (UAS7) on day 0, day 7, day 28, day 35 and day 56, and the Dermatology Life Quality Index (DLQI) on day 0, day 28, and day 56

SECONDARY OUTCOMES:
Improvement of sleep disturbance | Assessment of insomnia (common complications with urticaria) on starting day (day 0),day 28 and day 56
  Athens Insomnia Scale, Chinese edition (CAIS-8) is used to evaluate the improvement of sleep disturbance among chronic urticaria patient on day 0, day 28 and day 56
Changes of serologic markers for urticaria | Assessment of changes on serum markers for urticaria on starting day (day 0), day 28 and day 56
  Serum urticaria-related markers are checked on day 0, day 28 and day 56, including IgE, Eosinophil counts, CRP, IL-4, IL-6, IL-8, IL-10, IL-13, TNF-alpha and IFN-gamma

CONTACTS AND LOCATIONS:
Overall Officials: Sien-hung Yang, Ph.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Share data should be approved by the IRB before release

REFERENCES:
- [Background] Kato S, Kato TA, Nishie H, Nishima S, Iwanaga T, Monji A, Nakano M, Takeshita H, Furue M. Successful treatment of chronic urticaria with a Japanese herbal medicine, yokukansan. J Dermatol. 2010 Dec;37(12):1066-7. doi: 10.1111/j.1346-8138.2010.00937.x. Epub 2010 Sep 29. No abstract available. PMID 21083714
- [Background] Najib U, Bajwa ZH, Ostro MG, Sheikh J. A retrospective review of clinical presentation, thyroid autoimmunity, laboratory characteristics, and therapies used in patients with chronic idiopathic urticaria. Ann Allergy Asthma Immunol. 2009 Dec;103(6):496-501. doi: 10.1016/S1081-1206(10)60266-9. PMID 20084843
- [Background] Kulthanan K, Jiamton S, Thumpimukvatana N, Pinkaew S. Chronic idiopathic urticaria: prevalence and clinical course. J Dermatol. 2007 May;34(5):294-301. doi: 10.1111/j.1346-8138.2007.00276.x. PMID 17408437
- [Derived] Yang SH, Lin YH, Lin JR, Chen HY, Hu S, Yang YH, Yang YH, Yang YS, Fang YF. The Efficacy and Safety of a Fixed Combination of Chinese Herbal Medicine in Chronic Urticaria: A Randomized, Double-Blind, Placebo-Controlled Pilot Study. Front Pharmacol. 2018 Dec 18;9:1474. doi: 10.3389/fphar.2018.01474. eCollection 2018. PMID 30618764